CLINICAL TRIAL: NCT06495593
Title: Identifying Ocrelizumab-resistant Lymphocytes in Lymphoid Tissue in Multiple Sclerosis
Brief Title: Effects of Ocrelizumab Treatment on Immune Cells in Lymph Nodes in Multiple Sclerosis
Acronym: OCREFINA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ML45461
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Ocrelizumab; Lymph node; Lymphocyte
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RR-MS (Experimental): Two doses of 300 mg i.v. ocrelizumab two weeks apart followed by 600 mg i.v. ocrelizumab six months later.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Standard ocrelizumab dosing

SUMMARY:
B cell-depleting therapies, such as ocrelizumab, are among the most effective medications currently available for the treatment of multiple sclerosis (MS). This suggests that B cells play a very important role in MS. While B cells are rapidly eliminated from the blood of patients treated with medications like ocrelizumab, little is known about how effectively B cells are eliminated from lymph nodes, which are important sites of B cell activation. This study is being conducted to determine to what extent B cells are targeted in lymph nodes following ocrelizumab treatment, which may have important consequences for long-term MS outcomes.

DETAILED DESCRIPTION:
This is a phase IV single-arm observational study to study the effects of early ocrelizumab treatment on B cells and T cells in patients with multiple sclerosis (MS). Eligible patients must be 18-65 years old, have a diagnosis of relapsing-remitting MS, and have not been previously treated with a disease modifying therapy for MS, but plan to begin ocrelizumab treatment. Enrolled patients will undergo blood and lymph node fine needle aspiration before beginning treatment and again three months after treatment. Patients will receive two courses of ocrelizumab as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and be compliant with the study protocol
* The treating neurologist's independent medical assessment and decision to initiate the patient on ocrelizumab treatment as most appropriate standard of care for the patient
* Diagnosis of RR-MS with Expanded Disability Status Scale (EDSS) 0-5.5 at enrollment
* Treatment-naïve (i.e. no prior disease modifying therapy)
* Disease duration from the onset of MS symptoms: less than 15 years in patients with an EDSS greater than 5.0 at screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the treatment period and for 6 months after the final dose of ocrelizumab

Exclusion Criteria:

MS Related:

* Diagnosis of secondary progressive MS without relapses for at least 1 year.
* Diagnosis of primary progressive MS.
* Prior treatment with any disease modifying therapy for MS.
* Previous or concurrent treatment with any investigational agent or treatment with any experimental procedure for MS (e.g., treatment for chronic cerebrospinal venous insufficiency).

Infection Related:

* Known presence of recurrent or chronic infection (e.g., HIV, syphilis, tuberculosis).
* History of recurrent aspiration pneumonia requiring antibiotic therapy.
* History or known presence of infectious causes of myelopathy (e.g., syphilis, Lyme disease, HTLV-1, herpes zoster myelopathy).
* Known active bacterial, viral, fungal, mycobacterial infection, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infection of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks prior to baseline visit or oral antibiotics within 2 weeks prior to baseline visit.

Cancer Related:

- History of cancer, including solid tumors and hematological malignancies (except basal cell, in situ squamous cell carcinomas of the skin, and in situ carcinoma of the cervix or the uterus that have been excised and resolved with documented clean margins on pathology).

Women's health-related:

* Pregnant or lactating, or intending to become pregnant during the study
* Women of childbearing potential must have a negative serum or urine pregnancy test result within 14 days prior to initiation of study drug.

Other Medical Conditions:

* On systemic anti-coagulation or known blood clotting disorder.
* History of or currently active primary or secondary immunodeficiency.
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
* History of alcohol or other drug abuse within 24 weeks prior to enrollment.
* History or known presence of systemic autoimmune disorders, potentially causing progressive neurologic disease (e.g., lupus, anti-phospholipid antibody syndrome, Sjögren's syndrome, Behçet's disease).
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study.
* Significant, uncontrolled disease, as defined by AMA guidelines or similar, such as cardiovascular (including congestive heart failure - NYHA grade 3 or 4, cardiac arrhythmia), uncontrolled hypertension, pulmonary (including chronic obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus), gastrointestinal, or any other significant disease.
* Known presence or history of other neurologic disorders
* Systemic corticosteroid therapy within 4 weeks prior to baseline.
* Contraindications for, or intolerance to, oral or IV corticosteroids, including IV methylprednisolone, according to the country label, including hypersensitivity to any of the treatment drug constituents.
* Previous treatment with cyclophosphamide, mitoxantrone, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, total body irradiation, or bone marrow transplantation.

Laboratory:

* Positive serum or urine β-hCG.
* Positive for hepatitis B (hepatitis B surface antigen [HBsAg] positive or hepatitis B core antibody [total HBcAb] confirmed by positive viral DNA polymerase chain reaction [PCR]).
* AST or ALT more than 2 times the upper limit of normal.
* Platelet count below lower limit of normal.
* Total white blood cell count, including differential counts, below lower limit of normal.
* Absolute neutrophil count below lower limit of normal.
* Lymphocyte count below lower level of normal.
* Levels of serum IgG 18% below the lower limit of normal (LLN) and levels of serum IgM 8% below the LLN.
* Absolute CD4+ and CD8+ counts and CD4:CD8 ratio - within normal limits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Lymphocyte analysis | 3 months
  Percent reduction in B cells and T cell subsets in lymphoid tissue of MS patients following ocrelizumab treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sabatino, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No